CLINICAL TRIAL: NCT07311811
Title: An Open Label, Randomized, 2-sequence, 2-period, Fasting, Single Oral Dose, Crossover Study to Evaluate the Bioequivalence and Safety of 'IN-M00007' and 'IN-R00007' in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of IN-M00007 and IN-R00007 in Healthy Adult Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IN_RVZ_104
Record Dates: First submitted 2025-12-14; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): R → T R: IN-R00007, T: IN-M00007
  Interventions: Drug: IN-R00007; Drug: IN-M00007
- Sequence B (Experimental): T → R R: IN-R00007, T: IN-M00007
  Interventions: Drug: IN-R00007; Drug: IN-M00007

INTERVENTIONS:
Drug: IN-R00007 — Single dose
Drug: IN-M00007 — Single dose

SUMMARY:
This study aims to evaluate the Pharmacokinetic (PK) characteristics and safety after a single oral dose administration of IN-M00007 and IN-R00007 in healthy adult volunteers

DETAILED DESCRIPTION:
An open label, randomized, single oral dose, crossover study

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged ≥ 19 and < 60 years at screening
2. Body mass index(BMI) in the range of 18.0 and 30.0 kg/㎡

   * Body weight ≥ 50kg for male
   * Body weight ≥ 45kg for female
3. Subjects who do not have significant congenital or chronic diseases and without pathological symptoms or findings based on medical examinations(if necessary, EEG, ECG, chest X-ray, gastroscopy or gastrointestinal radiographic tests)
4. Determined by the investigator to be eligible for study participation based on the results of screening tests (e.g. hematology test, blood chemistry test, serology test, urinalysis, pregnancy diagnostic tests) conducted according to the IP characteristics
5. Subjects who voluntarily signed the consent form after receiving detailed explanation and understanding about purpose, details, characteristics of the IP and anticipated adverse events of the study
6. Subjects who agree to use highly effective methods of contraception(excluding hormonal methods) to preclude the possibility of pregnancy of themselves or their spouse/partner from the first IP administration until 14 days after the last administration, and who agrees not to donate sperm or ovum during this period

   * Highly effective contraceptive methods: intrauterine device(IUD), bilateral tubal ligation, a partner who has undergone vasectomy, or sexual abstinence However, periodic abstinence(calendar method, symptothermal method, post-ovulation method), withdrawal intercourse(coitus interruptus), spermicide methods, lactational amenorrhea method, and simultaneous use of female and male condoms are not considered contraceptive methods

Exclusion Criteria:

1. Subjects who have taken drugs which can induce(e.g, Barbiturates) or inhibit drug metabolism enzyme within 30 days prior to the start of the study(first IP administration day) or have taken medications that may affect this study within 10 days prior to the start of the study(first IP administration day)
2. Subjects who have participated in any other clinical study or bioequivalence study and administered IP within 6 months
3. Subjects who have donated whole blood within 8 weeks prior to the start of the study(first IP administration day) or have donated component blood within 2 weeks prior to the start of the study(first IP administration day)
4. Subjects with a history of gastrointestinal resection that may affect drug absorption(excluding appendectomy and hernia operation)
5. Subjects meeting following conditions within 1 month prior to the start of the study(first IP administration day)

   * Alcohol consumption > 21 glasses per week for male
   * Alcohol consumption > 14 glasses per week for female
6. Subjects with the following diseases

   * Subjects with hypersensitivity to the ingredient or components of this drug
   * Subjects with active liver disease or those with persistently elevated serum aminotransferase levels of unknown cause
   * Subjects with muscular disorders
   * Subjects receiving concomitant administration with cyclosporine
   * Subjects with severe renal impairment or kidney dysfunction
   * Subjects with a hereditary problems, for example, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
7. Subjects with a clinically significant history of mental illness
8. Pregnant or breastfeeding women if female
9. Subjects who are judged ineligible for the clinical study by the investigator due to reasons other than the above inclusion/exclusion criteria

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
PK parameter | Up to 48 hours
  AUCt of Rosuvastatin
PK parameter | Up to 48 hours
  Cmax of Rosuvastatin
PK parameter | Up to 72 hours
  AUCt of Ezetimibe
PK marameter | up to 72 hours
  Cmax of Ezetimibe

CONTACTS AND LOCATIONS:
Overall Officials: Hyeonggeon Kim, Principal Investigator — H Plus Yangji Hospital
Locations (1):
- H PLUS Yangji Hospital, Clinical Trial Center, Seoul, South Korea